CLINICAL TRIAL: NCT02857582
Title: Transplantation of Cultured Gut Microflora to Repeat Antibiotic-induced Diarrhea Due to Clostridium Difficile
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Per Hellström (Other)
Collaborators: Karolinska Institutet (Other); Region Gävleborg (Other)
Responsible Party: Sponsor-Investigator, Per Hellström, Professor, Uppsala University
Organization: Uppsala University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACHIM 1
Record Dates: First submitted 2016-07-26; First posted 2016-08-05 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Clostridium Difficile
Keywords: Antibiotic-induced diarrhea; Clostridium-difficile toxin; Pseudomembranous colitis
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Vancomycin; Metronidazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vancomycin (Active Comparator): Secondary treatment for relapse of Clostridium difficile infection.
  Interventions: Drug: Vancomycin; Drug: Metronidazole
- Cultured human intestinal microbiota1 (Experimental): Cultured intestinal microbiota is experimental treatment for relapse of Clostridium difficile infection.
  Interventions: Biological: Cultured human intestinal microbiota; Drug: Metronidazole
- Cultured human intestinal microbiota2 (Experimental): Cultured intestinal microbiota is thirdly experimental treatment for second relapse of Clostridium difficile infection.
  Interventions: Biological: Cultured human intestinal microbiota; Drug: Metronidazole

INTERVENTIONS:
Biological: Cultured human intestinal microbiota — Secondary treatment for C diff in replacement for regular vancomycin.
  Other Names: Anaerobic cultured human intestinal microbiota (ACHIM)
  Arms: Cultured human intestinal microbiota1; Cultured human intestinal microbiota2
Drug: Vancomycin — Active comparator to treatment with ACHIM
  Arms: Vancomycin
Drug: Metronidazole — Primary treatment for C diff in all treatment arms

SUMMARY:
Patients who have received antibiotics and thereafter developed diarrhea are investigated for presence of Clostridium difficile toxin. Primary treatment is given with oral metronidazole/vancomycin. In case of relapse, secondary treatment is given with either cultured gut microbiota rectally or oral vancomycin in sequence. In those cases where secondary treatment with vancomycin fails cultured gut microbiota is given as final treatment. As an extension treatment, all failures were treated with cluttered gut microbiota through the upper route. In both cases As an alternative cultured gut microbiota may be given via the duodenal route. Follow-up is carried out after 7, 30 and 90 days with interview and stool collection for analysis of Clostridium difficile.

ELIGIBILITY:
Inclusion Criteria:

* Antibiotic-induced diarrhea
* Positive fecal analysis for Clostridium difficile toxin

Exclusion Criteria:

* Antibiotic treatment
* Probiotic treatment
* Intestinal infection other than Clostridium difficile
* Inflammatory bowel disease (Ulcerative colitis, Crohn's disease
* Immunodeficiency (drug- och disease-related)
* Pregnancy
* Unable to accept endoscopic procedures
* Unable to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Normalization of stool consistency | 90 days
  Normalization according to Bristol stool scale

SECONDARY OUTCOMES:
Normalization of stool frequency | 90 days
  Normalization to less than three bowel movements per day

CONTACTS AND LOCATIONS:
Overall Officials: Hellström M Per, MD, PhD, Study Director — Uppsala University
Locations (1):
- Gävle Hospital, Gävle, Gävleborg County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Result] Bakken JS, Borody T, Brandt LJ, Brill JV, Demarco DC, Franzos MA, Kelly C, Khoruts A, Louie T, Martinelli LP, Moore TA, Russell G, Surawicz C; Fecal Microbiota Transplantation Workgroup. Treating Clostridium difficile infection with fecal microbiota transplantation. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1044-9. doi: 10.1016/j.cgh.2011.08.014. Epub 2011 Aug 24. PMID 21871249
- [Result] Husebye E, Hellstrom PM, Sundler F, Chen J, Midtvedt T. Influence of microbial species on small intestinal myoelectric activity and transit in germ-free rats. Am J Physiol Gastrointest Liver Physiol. 2001 Mar;280(3):G368-80. doi: 10.1152/ajpgi.2001.280.3.G368. PMID 11171619
- [Result] Gustafsson A, Berstad A, Lund-Tonnesen S, Midtvedt T, Norin E. The effect of faecal enema on five microflora-associated characteristics in patients with antibiotic-associated diarrhoea. Scand J Gastroenterol. 1999 Jun;34(6):580-6. doi: 10.1080/003655299750026038. PMID 10440607
- [Result] Gustafsson A, Lund-Tonnesen S, Berstad A, Midtvedt T, Norin E. Faecal short-chain fatty acids in patients with antibiotic-associated diarrhoea, before and after faecal enema treatment. Scand J Gastroenterol. 1998 Jul;33(7):721-7. doi: 10.1080/00365529850171666. PMID 9712236